CLINICAL TRIAL: NCT02778828
Title: Determination of Pharmacokinetic and Therapeutic Adaptation of Linezolid in the Treatment of Multi-Resistant Tuberculosis MDR-TB
Brief Title: Pharmacokinetic and Therapeutic Adaptation of Linezolid in the Treatment of Multi-Resistant Tuberculosis
Acronym: LINEZOLIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LINEZOLIDE
Record Dates: First submitted 2016-05-12; First posted 2016-05-20 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2018-08

CONDITIONS: Tuberculosis
Keywords: linezolide; tuberculosis; MDR-TB
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Multidrug-Resistant | interventions — Linezolid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients with Multi-Resistant Tb (Experimental)
  Interventions: Drug: Linezolid

INTERVENTIONS:
Drug: Linezolid — adjustment of Linezolid of based on the AUC/MIC and % T> MIC for each patient to confirm the appropriateness, in light of the peak and residual, and the interest of the split doses more frequently performed in case of too low residual or toxicity.

SUMMARY:
Linezolid, primary treatment for MDR-TB combination therapy anti. Until it is the dose of 600 mg x1 / day, rather sensible for most patients is more, which was unanimous. It is true that if a dosage is consensus, it goes without saying, because of the interindividual variability, marked moreover to linezolid, a therapeutic monitoring assay of plasma levels is indispensable for most pharmacological treatments. This therapeutic drug monitoring (TDM) often gives rise, as known, to dosage changes. It turns out that at present no real STP on the basic objectives PK / PD is really made in France in the treatment of tuberculosis (TB) and the bibliography remains rather poor recommendations, and yet all the elements are there: indeed linezolid is an antibiotic whose activity is purely "time-dependent". So one should fulfill 2 PK / PD objectives whose precise boundaries are sometimes still to be determined:

-% T> MIC, or percentage of time spent with plasma concentrations above the minimum inhibitory concentration of linezolid (LNZ) for Mycobacterium tuberculosis. In practice, the residual concentration before the next shot must be> MIC (0.125 to 1 mg / l)

* A fortiori it must also take into account the concentration preventing the appearance of resistant mutants, amounting to 1.2 mg / l
* AUC / MIC> 80, or ratio of the area under the curve (AUC, Area under curve) of plasma concentration versus time and CMI LNZ Until then, and without real bibliographic support, and for the sake of kindness to patients coupled with an economic advantage, the STP consisted of 2 samples, a peak 1:30 after taking (Cmax) and a residual before taking (C min) , after all, to 600mg x1 / 24 correlates well with the AUC (55% peak and 75% for the residual).

Following an observation that 25 to 30% of patients had a C min <1.2 mg / L, and even frequently <0.2 mg / L to 600 mg x 1, with some low peaks and leaving presage an AUC may be insufficient well.

This study is therefore more imperative to be a pharmacological streamlining and ensuring adequate therapeutic monitoring involves both maximum and minimum toxicity efficiency. And in the light of what has already been practiced for other molecules such as mycophenolate for example which is carried AUC or miniAUC for example. It would therefore be in the achievement of AUC in all patients treated with LNZ for TB MDR / XDR for over a week. Achieving this requires AUC obtaining 7 blood samples given day instead of two samples taken at present. Indeed one must have in mind that the peak of rational / residual has become blurred in this context, and that one of the two goals PK / PD is now filled (Cmin> MIC / CMP) but it should not be that not at the expense of the second (AUC). The benefits, direct and indirect are multiple and obtaining them is ensured through this protocol. The study by analyzing individual data will confirm the accuracy of the dose fractionation 300mgx2 / day and at a time to highlight a potential new dosage adjustment that would need to achieve for further study, so a substantial gain in terms of efficacy and toxicity via a suitable therapeutic monitoring. Secondly, determine which collection points, in these patients, these doses will be most interesting to take later in the routine of STP in order to collect less points (eg miniAUC MPA) retaining same statistical power to estimate kinetic parameters, mainly the AUC (eg aminoglycoside also). Finally in a third phase construction on the basis of these individual kinetics of a population pharmacokinetic model with highlighting of population parameters and especially co-related variables explaining the high pharmacokinetic variability and allowing for following patients to determine the individually tailored dose immediately before the first shot and the first assays.

DETAILED DESCRIPTION:
Primary objective :

Determination of the AUC / MIC and% T> MIC for each patient to confirm the appropriateness, in light of the peak and residual, and the interest of the split doses more frequently performed in case of too low residual toxicity or secondary objective: Determination of points of privileged samples in this context for maximum statistical power and minimal stress for the patient.

- Outlook: Development of a population PK model and determination of co-variables of interest and individualized dosages immediately for the next patients

Methodology :

Prospective, multi-center, non-interventional type of routine care Study duration: 1 day / patient, maximum total duration of recruitment: 6 months, aim 30-40patients included

Acquisition of data:

Additional media (Informed consent, sampling protocol, collection form of biological, clinical and pharmacological patient and treatment)

* Statistical analysis by a software suitable pharmacokinetic
* Anonymity of data: an identifier for each subject will be awarded (first name and surname / number) and the data will be entered in a computer file that will be retained by the sponsor on the GHPSJ site for the realization of determinations of AUC and optimal dosages.

Development of the study:

* Performance of the study
* Expected duration of patient recruitment: up to 6 months
* Number of patients to recruit 30 to 40 patients, limited by the number of hospitalized patients in the recruiting center (sanatorium Bligny), combining both MDR-TB and treatment with linezolid
* Duration of the study for each patient: 12 to 24 hours the time for the 7 samples.
* Regarding the iterative sampling and prevention of potentially associated pain, most patients already have a KT or a PAC in place for administering IV drugs (amiklin, augmentin or vitamins in particular), it is therefore on these it is planned to take samples. For the few patients with no system in place for use, it will be explained and proposed the establishment of a device Catelon and a patch Emla, the decision on the matter will be up to the patient.

Destruction of samples: the samples will not be retained after being used for the study. They will be destroyed in accordance with the rules of good practice research laboratories.

Data: Data include clinical and biological, bacteriological patient. The GHPSJ guarantee that the biological material will be digitally encoded and will not involve direct identifying information of subjects participating in research. The shipment will be made by the sanatorium Bligny staff under the supervision of the investigator within the department (Dr Mathilde Jachym and Damien Le Du).

Ethical aspects: After notification of the CPP Ile de France II, the project will be classified as "research in routine care." The opinion of the CPP Ile de France II will be requested at the meeting of June 2015. The manager research center will be the hospital group Paris Saint-Joseph (GHPSJ). The latter will contract with the SHAM (usual insurer GHPSJ for care and clinical research) to ensure the risk of the blood sample.

The research information will be issued and the signature of the Circular will be collected from the patient. An agreement will be made between institutions, and the GHPSJ Bligny Medical Center, including the logistics of transport and harvest management.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* MDR-TB / XDR
* Treated by Linezolide per os at total daily dose of 600 mg-treatment started for> 7 days
* BMI <35 kg / m²

Exclusion Criteria:

* Age <18 years
* Treatment By Linezolide PO at a dose> or <600mg / d or I.V.
* Treatment Started since <7 days (Plock, 2007)
* Insufficient moderate renal or severe / dialysis
* BMI> 35 kg / m²

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-11-04 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Air Under the Curve (AUC) of Linezolid concentration | 30 minutes after oral intaking linezolid
Minimum Inhibitory Concentration (MIC) of Linezolid | 30 minutes after oral intaking linezolid

CONTACTS AND LOCATIONS:
Overall Officials: Alban LE MONNIER, MD, Principal Investigator — Groupe Hospitalier Paris Saint-Joseph (FRANCE)
Locations (1):
- Sanatorium du Petit Fontainebleau Centre Médical de Bligny, Briis-sous-Forges, Essonne, France

IPD SHARING:
Plan to Share IPD: Undecided